CLINICAL TRIAL: NCT04815876
Title: Randomized Trial Comparing Transperineal vs. Transrectal MRI-targeted Prostate Biopsy; Randomized Controlled Trial Assessing Transperineal Prostate Biopsy to Reduce Infection Complications
Brief Title: PReclude Infection EVEnts With No Prophylaxis Transperineal Biopsy 2
Acronym: PREVENT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21-03023431; CER-2019C2-17372 (Other: Patient-Centered Outcomes Research Institute); 18-02-365-PCORI (Other: Biomedical Research Alliance of New York (BRANY))
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Infection
Keywords: prostate cancer; prostate biopsy; biopsy infection; fusion biopsy; MRI-targeted biopsy; transperineal; transrectal
MeSH Terms: conditions — Infections; Prostatic Neoplasms | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Men enrolled in this prospective, randomized trial will be randomized in a 1:1 ratio to receive either transperineal MRI-targeted or transrectal MRI-targeted prostate biopsy.
Who Masked: Outcomes Assessor
Masking Description: Radiologists assessing MRI results are blinded to treatment assignment. Pathologists assessing biopsy results are blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transrectal (Active Comparator): Patients will receive a transrectal MRI-guided prostate biopsy.
  Interventions: Procedure: Transrectal MRI-guided prostate biopsy; Drug: Antibiotic (prophylaxis)
- Transperineal (Active Comparator): Patients will receive a transperineal MRI-guided prostate biopsy.
  Interventions: Procedure: Transperineal MRI-guided prostate biopsy

INTERVENTIONS:
Procedure: Transperineal MRI-guided prostate biopsy — Transperineal prostate biopsy will be performed under local anesthesia in the office. This approach avoids transrectal needle tracking.
  Arms: Transperineal
Procedure: Transrectal MRI-guided prostate biopsy — Transrectal prostate biopsy is currently the most popular approach to evaluate a positive screening test for prostate cancer.
  Arms: Transrectal
Drug: Antibiotic (prophylaxis) — For men undergoing transrectal biopsy, antibiotic prophylaxis will be administered in accordance with guidelines from the American Urological Association (AUA).
  No antibiotic prophylaxis will be administered for men undergoing transperineal biopsy.
  Arms: Transrectal

SUMMARY:
Approximately one million transrectal prostate biopsies are performed annually in the U.S., and the risk of post- biopsy infection is increasing due to greater antibiotic resistance of rectal flora. Preliminary data demonstrates that a transperineal MRI-targeted biopsy approach under local anesthesia compared to the standard practice transrectal MRI-targeted prostate biopsy has a much lower risk of infection, comparable pain/discomfort and may improve detection of prostate cancer.

This randomized controlled trial will be the first prospective study to evaluate in-office transperineal MRI targeted prostate biopsy.

The investigators hypothesize that a transperineal MRI-targeted biopsy approach under local anesthesia compared to the standard practice transrectal MRI-targeted prostate biopsy has a much lower risk of infection, comparable pain/discomfort and may improve detection of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the most commonly diagnosed malignancy in U.S. men. There are approximately 1 million prostate biopsy performed annually in the U.S. Almost all biopsies are performed as an office based procedure in under 15 minutes. The precision of biopsy has improved over the last decade with the introduction of MRI guidance/targeting of suspicious lesions within the prostate.

However, significant limitations remain with this approach, including a significantly increasing risk of post-biopsy infection. This arises because more than 97% of all prostate biopsy are performed via a transrectal approach that introduces rectal bacteria with each pass of the biopsy needle into the sterile urinary tract. The current risk of post-transrectal biopsy infection, even with antimicrobial prophylaxis, is high at approximately 7% overall with 3% (30,000 men) requiring hospitalization annually.

Transperineal biopsy is an alternate approach that eliminates the direct introduction of bacteria from the rectum to the prostate. This approach, which is performed without antimicrobial prophylaxis, instead passes the biopsy needle through the perineal skin and pelvic floor.

Transperineal biopsy has not been widely adopted for several reasons. Historically, it has been considered too painful for patients in the clinic and thus was traditionally performed under general anesthesia. The added time, inconvenience and cost has limited its national adoptance. Second, when transrectal biopsy was initially adopted over 40 years ago, antibiotic resistance of rectal flora was not a challenge.

Beyond the potential for in-office transperineal biopsy to significantly reduce or eliminate biopsy infections, transperineal biopsy may also improve cancer detection: studies of transperineal biopsy (performed under general anesthesia) demonstrate higher detection rates for prostate cancer, particularly for anterior zone tumors, compared to transrectal biopsy. This is notable, as anterior tumors are difficult to sample with transrectal. Anterior tumors are also twice as likely to occur in African American men. In fact, our research demonstrates that some of the outcomes disparities in African American men may stem from an underdiagnosis of anterior prostate cancers.

Although transrectal biopsy is used widely, it is associated with a significant and increasing risk of biopsy infections due to growing antibiotic resistance, highlighting the urgent need for a safer alternative approach to prostate biopsy. The study investigators have refined a transperineal approach under local anesthesia with MRI-targeting/guidance without the need for antibiotic prophylaxis. The investigators hypothesize that transperineal MRI targeted biopsy will: (1) largely eliminate post-biopsy infections and costly hospitalizations for urosepsis; (2) be performed in the office with similar discomfort and non-infectious complications compared to transrectal MRI targeted biopsy; and (3) have significantly better detection of prostate cancer.

This multi-center randomized controlled trial will be conducted to evaluate in-office transperineal MRI targeted vs. transrectal MRI targeted biopsy, the current gold standard. This has transformative impact to change current standard of practice.

ELIGIBILITY:
Inclusion Criteria:

* Active surveillance cohort: History of Grade Group 1 prostate cancer, first diagnosed ≤24 months prior to date of planned confirmatory biopsy and diagnostic biopsy was preceded by a multiparametric MRI of the prostate
* Prior negative cohort: Clinical concern for the presence of prostate cancer as determined by the treating urologist and prior negative prostate biopsy performed ≤36 months prior to date of planned biopsy
* Willingness to sign informed consent and adhere to the study protocol

Exclusion Criteria:

* Acute prostatitis within the last 6 months
* Current non-urologic bacterial infection requiring active treatment with antibiotics
* Unfit to undergo prostate biopsy under local anesthesia
* Prior definitive therapy for prostate cancer, such as radiation therapy or partial gland ablation
* Contraindication to prostate MRI (claustrophobia, pacemaker, chronic kidney disease)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1302 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in infection adverse events, as measured on TRUS-BxQ | At initiation of biopsy, immediately following biopsy, 7 days post-biopsy
  TRUS-BxQ is a validated biopsy questionnaire that measures adverse events that have occurred due to infection. Patient questionnaire consists of Yes/No questions about infection complications and duration of infection.

SECONDARY OUTCOMES:
Change in patient-reported pain and discomfort, as measured on a 0-10 Likert scale | Immediately following biopsy, 7 days post-biopsy
  Pain and discomfort will be scored on a 0-10 Likert scale. 0 indicates no pain/discomfort and high scores indicate greater pain/discomfort.
Change in patient-reported anxiety, as measured on a 0-10 Likert scale | Immediately following biopsy, 7 days post-biopsy
  Anxiety will be scored on a 0-10 Likert scale. 0 indicates no anxiety and high scores indicate greater anxiety.
Detection of clinically significant disease as measured by Gleason Grade Group ≥ 2 | 7 days post-biopsy
  Gleason Grade Group is a prostate cancer grading system released by the International Society of Urological Pathology (ISUP). Grade Group 1 indicates Low/Very Low Risk, Grade Group 2 indicates Intermediate (Favorable) Risk, Grade Group 3 indicates Intermediate (Unfavorable) Risk, and Grade Groups 4 and 5 indicate High/Very High Risk.
  Prostate cancer grade will be categorized into insignificant (Gleason Grade Group 1) and clinically significant (Grade Group ≥ 2).
Change in adverse events, as measured on TRUS-BxQ | At initiation of biopsy, immediately following biopsy, 7 days post-biopsy
  TRUS-BxQ is a validated biopsy questionnaire that measures adverse events that have occurred, such as hospital re-admissions, aborted procedures due to discomfort, hematuria, urinary retention, hematospermia, and/or hematochezia. Patient questionnaire consists of Yes/No questions about general complications and duration of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Hu, MD MPH, Principal Investigator — Weill Cornell Medicine, NewYork-Presbyterian
Locations (16):
- United States (16):
  - University of Southern California, Los Angeles, California
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - NewYork-Presbyterian Queens, Flushing, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Einstein Healthcare Network, Elkins Park, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplan-Marans E, Zhang TR, Hu JC. Differing Recommendations on Prostate Biopsy Approach to Minimize Infections: An Examination of the European Association of Urology and American Urological Association Guidelines. Eur Urol. 2023 Nov;84(5):445-446. doi: 10.1016/j.eururo.2023.05.036. Epub 2023 Jun 7. PMID 37296040
- [Derived] Hu J, Zhu A, Vickers A, Allaf ME, Ehdaie B, Schaeffer A, Pavlovich C, Ross AE, Green DA, Wang G, Ginzburg S, Montgomery JS, George A, Graham JN, Ristau BT, Correa A, Shoag JE, Kowalczyk KJ, Zhang TR, Schaeffer EM. Protocol of a multicentre randomised controlled trial assessing transperineal prostate biopsy to reduce infectiouscomplications. BMJ Open. 2023 May 19;13(5):e071191. doi: 10.1136/bmjopen-2022-071191. PMID 37208135